CLINICAL TRIAL: NCT04068051
Title: An Open-Label, Long-Term Study to Assess the Safety and Efficacy of AXS-07 (MoSEIC™ Meloxicam and Rizatriptan) for the Acute Treatment of Migraine in Adults
Brief Title: Multimechanistic Treatment Over Time of Migraine Symptoms (MOVEMENT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AXS-07-302
Record Dates: First submitted 2019-07-27; First posted 2019-08-28 (Actual); Results first posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Migraine
Keywords: Axsome; AXS-07; MoSEIC™ meloxicam; rizatriptan
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AXS-07 (Experimental)
  Interventions: Drug: AXS-07

INTERVENTIONS:
Drug: AXS-07 — AXS-07 (MoSEIC meloxicam and rizatriptan) taken by mouth for the acute treatment of migraine.

SUMMARY:
MOVEMENT (Multimechanistic Treatment over Time of Migraine Symptoms) is a Phase 3 study to evaluate the long-term safety of chronic intermittent use of AXS-07 and to assess the effect of AXS-07 on migraine symptoms following repeated treatment of migraine attacks.

DETAILED DESCRIPTION:
This study is a Phase 3, multicenter, open-label, trial to evaluate the long-term safety and efficacy of intermittent chronic dosing with AXS-07 in subjects with migraine attacks. Eligible subjects will take AXS-07 following the onset of a migraine. Subjects will be treated for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Has participated in a prior study with AXS-07 for the treatment of migraine

Exclusion Criteria:

* Has previously received any investigational drug or device or investigational therapy within 30 days before Screening, other than AXS-07
* Pregnant, breastfeeding, or planning to become pregnant or breastfeed during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 706 (Actual)
Dates: Start 2019-07-06 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (49):
- United States (49):
  - Clinical Research Site, Birmingham, Alabama
  - Clinical Research Site, Mobile, Alabama
  - Clinical Research Site, Phoenix, Arizona
  - Clinical Research Site, Canoga Park, California
  - Clinical Research Site, Colton, California
  - Clinical Research Site, Encino, California
  - Clinical Research Site, Los Alamitos, California
  - Clinical Research Site, Los Angeles, California
  - Clinical Research Site, San Diego, California
  - Clinical Research Site, Spring Valley, California
  - Clinical Research Site, Walnut Creek, California
  - Clinical Research Site, Hallandale, Florida
  - Clinical Research Site, Jacksonville, Florida
  - Clinical Research Site, Lake City, Florida
  - Clinical Research Site, Lake Worth, Florida
  - Clinical Research Site, Miami, Florida
  - Clinical Research Site, Ocoee, Florida
  - Clinical Research Site, Orlando, Florida
  - Clinical Research Site, Ormond Beach, Florida
  - Clinical Research Site, Tampa, Florida
  - Clinical Research Site, Stockbridge, Georgia
  - Clinical Research Site, Evanston, Illinois
  - Clinical Research Site, Louisville, Kentucky
  - Clinical Research Site, Boston, Massachusetts
  - Clinical Research Site, North Dartmouth, Massachusetts
  - Clinical Research Site, Waltham, Massachusetts
  - Clinical Research Site, Ann Arbor, Michigan
  - Clinical Research Site, Minneapolis, Minnesota
  - Clinical Research Site, Springfield, Missouri
  - Clinical Research Site, Las Vegas, Nevada
  - Clinical Research Site, Albuquerque, New Mexico
  - Clinical Research Site, Manlius, New York
  - Clinical Research Site, Rochester, New York
  - Clinical Research Site, Williamsville, New York
  - Clinical Research Site, High Point, North Carolina
  - Clinical Research Site, Cincinnati, Ohio
  - Clinical Research Site, Columbus, Ohio
  - Clinical Research Site, Oklahoma City, Oklahoma
  - Clinical Research Site, Portland, Oregon
  - Clinical Research Site, Salem, Oregon
  - Clinical Research Site, Philadelphia, Pennsylvania
  - Clinical Research Site, Charleston, South Carolina
  - Clinical Research Site, Mt. Pleasant, South Carolina
  - Clinical Research Site, Knoxville, Tennessee
  - Clinical Research Site, Memphis, Tennessee
  - Clinical Research Site, Austin, Texas
  - Clinical Research Site, Salt Lake City, Utah
  - Clinical Research Site, Charlottesville, Virginia
  - Clinical Research Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AXS-07: AXS-07 (MoSEIC™ meloxicam and rizatriptan) taken by mouth for the acute treatment of migraine.
Period: Overall Study
Arm/Group | AXS-07
Started | 706
Completed | 138
Not Completed | 568

BASELINE CHARACTERISTICS:
Population: Safety Population includes all subjects who received at least one dose of study drug.
Arm/Group | AXS-07
Number analyzed (Participants) | 706
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (10.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 580
  Male | 126
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 132
  White | 544
  More than one race | 9
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Long-term Safety of Chronic Intermittent Use of AXS-07
Description: Long-term safety as measured by:
  Subjects with any TEAEs
  Subjects with suspected to be drug-related TEAEs
  Subjects with serious TEAEs
  Subjects with TEAEs that led to drug withdrawal
  Subjects with TEAEs that led to withdrawal from study
  Subjects with TEAEs that resulted in death
Time Frame: Up to 12 months
Population: Safety Population includes all subjects who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | AXS-07
Number analyzed (Participants) | 706
Participants
  Subjects with any TEAEs | 293
  Subjects with suspected to be drug-related TEAEs | 118
  Subjects with serious TEAEs | 8
  Subjects with TEAEs that led to drug withdrawal | 10
  Subjects with TEAEs that led to withdrawal from study | 13
  Subjects with TEAEs that resulted in death | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected after administration of study drug through the final visit (up to 12 months). Any AE was monitored up to a maximum of 30 days after the final visit.
Description: Safety Population includes all subjects who received at least one dose of study drug.
Arm/Group | AXS-07
All-Cause Mortality (participants affected / at risk) | 0/706
Serious Adverse Events (participants affected / at risk) | 8/706
Other Adverse Events (participants affected / at risk) | 95/706
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXS-07 (N=706)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 1 (1)
Burns third degree (Injury, poisoning and procedural complications) | 1 (1)
Musculoskeletal procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1)
Victim of crime (Social circumstances) | 1 (1)
Skin graft (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXS-07 (N=706)
Nausea (Gastrointestinal disorders) | 40 (88)
Vomiting (Gastrointestinal disorders) | 33 (48)
Dizziness (Nervous system disorders) | 22 (45)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-17): https://cdn.clinicaltrials.gov/large-docs/51/NCT04068051/Prot_SAP_000.pdf